CLINICAL TRIAL: NCT01206777
Title: Assessment of Hypersensitivity Reactions and Feasibility of a 60 Minute Rapid Infusion Rituximab Protocol in Patients With B-Cell Non-Hodgkin's Lymphoma (NHL) and Chronic Lymphocytic Leukemia (CLL) at a Comprehensive Cancer Center
Brief Title: Feasibility Study of a 60 Minute Rapid Infusion Rituximab Protocol in Patients With B-cell Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-10001; NCI-2012-00929 (Registry Identifier: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2010-09-10; First posted 2010-09-22 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Indolent or Intermediate Grade B-cell Malignancy
Keywords: Hypersensitivity Reactions; B-cell malignancies
MeSH Terms: conditions — Hypersensitivity | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab (Experimental)
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Dose 2 of Rituximab IVPB will be started at a rate of 100 mg/hr for the first 15 minutes. If tolerated, the remainder of the bag will be infused over 45 minutes.

SUMMARY:
The purpose of this study is to assess the feasibility of a 60 minute rapid infusion rituximab protocol in the institution's outpatient infusion center.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-89
* Diagnosis of indolent or intermediate grade B-cell malignancy
* Patients receiving rituximab-based therapy at a dose of 375mg/m2, regardless of weight
* First dose given within 3 months of the second dose
* Infusion scheduled for outpatient administration at The Arthur G. James Cancer Hospital and Richard J. Solove Research Institute

Exclusion Criteria:

* Diagnosis of aggressive lymphoma
* Absolute lymphocyte count > 10 x 103 cells/µL
* New York Heart Association (NYHA) classification Grade II or greater congestive heart failure
* Enrolled on another clinical trial
* Allergy to murine-containing medications
* Grade III or IV hypersensitivity reaction during the initial infusion of rituximab
* Prisoners
* Pregnant women
* Mentally or physically unable to give consent

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Jones, M.D., M.P.H., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Dotson E, Crawford B, Phillips G, Jones J. Sixty-minute infusion rituximab protocol allows for safe and efficient workflow. Support Care Cancer. 2016 Mar;24(3):1125-9. doi: 10.1007/s00520-015-2869-4. Epub 2015 Aug 14. PMID 26268782
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from October 2010 to April 2013
Period: Overall Study
Arm/Group | Rituximab
Started | 52
Discontinued Trial and Deemed Ineligible | 2
Completed | 50
Not Completed | 2
Not completed — Death | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab
Number analyzed (Participants) | 52
Age, Continuous [Median (Full Range); unit: years] | 63 [19 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 21
Region of Enrollment [Number; unit: patients]
  United States | 52

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Grade III and IV Hypersensitivity Reactions
Time Frame: Every 15 minutes from start of infusion until completion, for up to 1 hour
Measure: Number; unit: percentage of patients
Arm/Group | Rituximab
Number analyzed (Participants) | 50
percentage of patients | 0

2. Secondary Outcome: Time Savings of a 60 Minute Infusion Versus Predicted Infusion Time Using Standard Second Dose Titration Schedule
Time Frame: Determined from difference in expected time by package insert administration and actual time on day of treatment
Measure: Mean (95% Confidence Interval); unit: minutes for rapid R infusion
Arm/Group | Rituximab
Number analyzed (Participants) | 50
minutes for rapid R infusion | 62.4 [61.2 to 63.6]

3. Secondary Outcome: Demonstrate Nursing Satisfaction for Administration of Rapid Infusion Over Standard Titration Practice
Description: Surveys were given to nurses in the outpatient infusion center to measure their satisfaction with the administration of the rapid infusion rate compared to standard titration practice.
Time Frame: 6 months, as a before and after infusion survey
Population: Post infusion surveys were collected and de-identified by assignment of an individual nurse identification number
Measure: Number; unit: percentage of nurses satisfied
Arm/Group | Rituximab
Number analyzed (Participants) | 50
percentage of nurses satisfied | 100

ADVERSE EVENTS:
Description: The study utilized the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 for adverse event reporting.
Arm/Group | Rituximab
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes